CLINICAL TRIAL: NCT01743352
Title: Protocole ULTRAFAST - ECHOTRACKING : Remodelage pariétal et rigidité artérielle Chez l'Hypertendu : Nouvelle étude de Leur Relation Utilisant l'élastographie Par Ultrafast-écho et la séparation Intima/média Par écho-tracking
Brief Title: Comparison of Ultrafast Echo With Echotracking
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 2012-01; ID - RCB 2012-A01255-38 (Other: ANSM)
Record Dates: First submitted 2012-12-04; First posted 2012-12-06 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Essential Untreated Hypertension; Healthy Volunteers
Keywords: Large arteries; stiffness; intima media thickness; ultrasound imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hypertension patients: Local common carotid artery pulse wave velocity is compared in patients with hypertension and healthy volunteers.
- Healthy Volunteers: Local common carotid artery pulse wave velocity is compared in hypertension patients and healthy volunteers

SUMMARY:
The aim is to compare a new technique for assessing mechanical properties of large arteries: the Ultrafast echo with the reference technique, the echotracking. This will be done by studying in parallel hypertensive patients and controls with both techniques and this will revisit old concepts of increased stiffness in hypertensive arteries.

DETAILED DESCRIPTION:
Ultrafast ECHO is a new non invasive method for assessing stiffness of living tissues. It takes advantage of very fast imaging technologies (up to 20 000 images/sec) to measure the diffusion of pressure waves in the tissues. This pressure wave can be either natural (blood pressure), or generated by an very short ultrasonic impulsion at a given place. By using both modes, it is possible to have a precise cartography of tissue mechanical properties. This technique is applied to solid tissues such as breast or liver, but not yet currently to hollow tissues such as arteries. The aim of the present study is to compare the values of stiffness obtained with Ultrafast ECHO with the reference non invasive technique, the Echotracking, which measures stiffness by assessing the deformation of arteries in response to changes in blood pressure. On the physiological part, we will revisit old concepts of increased stiffness of hypertensive's arteries. Indeed, hypertension is associated with increased stiffness due to recruitement of collagen fibers, but also to chronic remodelling. We have shown before that this remodelling conducts to accumulation of arterial tissue of lesser intrinsic stiffness. The latter finding was done through models based on echotracking measurements. It will be interesting to see whether it holds true when stiffness is directly measured.

Sixty subjects (30 normotensive and30 hypertensives) will be included and studied once. Measurement will be performed in random order 3 time on the common carotid artery on both sides. Aortic stiffness will be measured by pulse wave velocity

ELIGIBILITY:
Inclusion Criteria:

* hypertension,
* essential (WHO workup),
* untreated (> 28 days of treatment interruption, < 6 months of treatment) on insufficiently equilibrated (BP > 140 and/or 90 mmHg)

Exclusion Criteria:

* Any concomitant severe disease compromising patient's participation or compliance

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting Essential untreated hypertension Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Local common carotid artery pulse wave velocity | Day 1

SECONDARY OUTCOMES:
Common carotid artery Young's modulus (Stiffness of wall material) | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Laurent, MD, PhD, Principal Investigator — Pharmacology Department - Hopital Européen Georges Pompidou - Paris
Locations (1):
- Hopital Européen Georges Pompidou / Service de Pharmacologie, Paris, France